CLINICAL TRIAL: NCT04144049
Title: A Randomized, Double-blind, Placebo-controlled, Dose Ranging, Parallel, Multi-center, Phase II Study to Evaluate the Efficacy and Safety of MT921 in Subjects With Moderate to Severe Submental Fat
Brief Title: A Phase II Study to Evaluate the Efficacy and Safety of MT921 in Subjects With Moderate to Severe Submental Fat
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MT11-KR18SMF203
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Submental Fat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MT921 (Experimental): 1% or 1.5%, subcutaneously administered at most 50 injections per treatment.
  Interventions: Drug: MT921
- Placebo (Placebo Comparator): Subcutaneously administered at most 50 injections per treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT921 — Subcutaneously administered, 0.2ml per injection, at most 50 injections per treatment session.
  Arms: MT921
Drug: Placebo — Subcutaneously administered, 0.2ml per injection, at most 50 injections per treatment session.
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, dose-ranging, parallel, multi-center, phase II study to evaluate the efficacy and safety of MT921 in subjects with moderate to severe submental fat.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 19 and under 65 years old
* Subjects achieving CA-SMFRS and PA-SMFRS score of 2 or 3
* Subjects who voluntarily signed the Informed Consent

Exclusion Criteria:

* Subjects who had liposuction or other procedures on the treatment area that might affect the assessment.
* Subjects with BMI over 35.0kg/m^2
* Subjects with dysphagia
* Subjects who are allergic or hypersensitive to the investigational product
* Subjects who are pregnant or lactating, or does not agree to use an accepatble form of contraception during the clinical trial.
* Subjects who are otherwise deemed uneligible by the investigator.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
Responder rate of 2-grade improvement in CA-SMFRS | 4 weeks after the last treatment session
  Proportion of subjects who have at least a 2-grade improvement from basleine on the Clinician Assessed-SubMental Fat Rating Scale (5-point scale, 0-No submental fat to 4-Excessive submental fat) at 4 weeks after the last treatment.
Responder rate of 2-grade improvement in PA-SMFRS | 4 weeks after the last treatment session
  Proportion of subjects who have at least a 2-grade improvement from basleine on the Patient Assessed-SubMental Fat Rating Scale (5-point scale, 0-No submental fat to 4-Excessive submental fat) at 4 weeks after the last treatment.
Responder rate of 1-grade improvement in CA-SMFRS | 4 weeks after the last treatment session
  Proportion of subjects who have at least a 1-grade improvement from basleine on the Clinician Assessed-SubMental Fat Rating Scale (5-point scale, 0-No submental fat to 4-Excessive submental fat) at 4 weeks after the last treatment.
Responder rate of 1-grade improvement in PA-SMFRS | 4 weeks after the last treatment session
  Proportion of subjects who have at least a 1-grade improvement from basleine on the Patient Assessed-SubMental Fat Rating Scale (5-point scale, 0-No submental fat to 4-Excessive submental fat) at 4 weeks after the last treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-ang University Hospital, Seoul, South Korea